CLINICAL TRIAL: NCT00407004
Title: Effect of Extracorporeal Liver Support by MARS and Prometheus on Albumin-Bound Substances in Acute-on-Chronic Liver Failure
Brief Title: Elimination of Albumin-Bound Substances by MARS and Prometheus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EAT
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Liver Failure
Keywords: acute-on-chronic liver failure, MARS, Prometheus, bilirubin, bile acids, cytokines
MeSH Terms: conditions — Liver Failure; Acute-On-Chronic Liver Failure

INTERVENTIONS:
Device: MARS (Molecular Adsorbents Recirculating System)
Device: Prometheus (FPSA, Fractionated Plasma Separation and Adsorption)

SUMMARY:
This trial compares the efficacy of two artificial liver support systems, MARS (Molecular Adsorbents Recirculating System) and Prometheus (FPSA, Fractionated Plasma Separation and Adsorption), in removing albumin-bound substances such as bilirubin, bile acids, and cytokines.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with acute-on-chronic liver failure (severe deterioration of chronic liver disease) unresponsive to standard medical treatment for >=48 hours

Exclusion Criteria:

* arterial hypotension
* extrahepatic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-03; Study Completion 2004-04

PRIMARY OUTCOMES:
serum levels of albumin-bound substances

SECONDARY OUTCOMES:
plasma clearance of albumin-bound substances

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf E. Stauber, MD, Principal Investigator — Medical University of Graz; Peter Krisper, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Result] Krisper P, Haditsch B, Stauber R, Jung A, Stadlbauer V, Trauner M, Holzer H, Schneditz D. In vivo quantification of liver dialysis: comparison of albumin dialysis and fractionated plasma separation. J Hepatol. 2005 Sep;43(3):451-7. doi: 10.1016/j.jhep.2005.02.038. PMID 16023249
- [Result] Jung A, Krisper P, Haditsch B, Stauber RE, Trauner M, Holzer H, Schneditz D. Bilirubin kinetic modeling for quantification of extracorporeal liver support. Blood Purif. 2006;24(4):413-22. doi: 10.1159/000094575. Epub 2006 Jul 14. PMID 16847391